CLINICAL TRIAL: NCT03414853
Title: Prospective Study of a Free-text Diagnosis Prediction Algorithm for Appendicitis in the Emergency Department
Brief Title: Free Text Prediction Algorithm for Appendicitis
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: N-171-000-456-001
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Acute Appendicitis; Abdominal Pain
Keywords: Appendicitis, abdominal pain, free text prediction
MeSH Terms: conditions — Appendicitis; Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With algorithm use
  Interventions: Diagnostic Test: Free text prediction algorithm for appendicitis
- No algorithm use

INTERVENTIONS:
Diagnostic Test: Free text prediction algorithm for appendicitis — A free-text prediction software that predicts the probability of acute appendicitis
  Groups: With algorithm use

SUMMARY:
Computer-aided diagnostic software has been used to assist physicians in various ways. Text-based prediction algorithms have been trained on past medical records through data mining and feature analysis. Currently, all text-based machine learning prediction problem models have been built on extracted data with no research completed on free text based prediction algorithms. This study aims to determine the accuracy of a free text prediction algorithm in predicting the probability of appendicitis in patients presenting to the Emergency Department with abdominal pain and gastrointestinal symptoms.

DETAILED DESCRIPTION:
Developing machine learning models that have a strong prediction power for diagnosis of appendicitis from physician entered free text input can improve diagnostic accuracy of doctors. It also offers the possibility of using prediction algorithms to improve routine clinical care. In the future, multiple machine learning models can be combined to increase prediction accuracy and prediction algorithms can be extended to other diagnoses.

18,000 cases of emergency department presentations over 10 years were used as a training and validation dataset. To develop the appendicitis prediction model, deep learning neural networks with a customized medical ontology were used. The diagnostic accuracy of the model is expressed as sensitivity (recall), specificity and F1 score (harmonic mean). The developed diagnosis predictive model shows high sensitivity (86.3%), specificity (91.9%) and F1 score (88.8) in diagnosing appendicitis from patients presenting with abdominal pain.

The predictive model algorithm will also highlight words in the free text (entered by the attending physician) that it assigns higher probability for predicting an outcome. The doctors will be instructed to provide a percentage likelihood of appendicitis based on the clinical presentation and any available laboratory investigations. The doctor is then shown the prediction of the algorithm as well as the highlighted words for the patient entered. He/she must then provide another prediction of the likelihood of appendicitis after seeing the algorithm generated prediction.

The aim is to evaluate the performance of the algorithm and to assess if usage of the algorithm is able to help emergency doctors improve their diagnosis of appendicitis. The prediction results will be tabulated to assess accuracy of the algorithm, doctors before algorithm input and doctors after receiving algorithm input. The accuracy will be expressed as sensitivity, specificity, accuracy, positive prediction value, F1 score and F0.5 score.

Approximately 100 emergency doctors will be recruited over the course of 1 year as participants in the study. The doctors will be split randomly assigned to two groups - the algorithm arm and the no algorithm arm. The randomization will be by time (weekly) using variable block randomization of 4 and 6. The patients will be followed up for the final discharge diagnoses.

ELIGIBILITY:
Eligibility criteria of doctors- Inclusion criteria: Junior doctors working in the Emergency Department Exclusion criteria: Refusal of consent

Eligibility criteria of patients-

Inclusion Criteria:

* Presence of abdominal pain, OR
* Presence of gastrointestinal symptoms such as nausea, vomiting or diarrhea, OR
* Fever with anorexia

Exclusion Criteria:

* Previous history of appendicectomy
* Refusal of consent

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Attending physicians will be recruited as study participants and randomised weekly into "algorithm use" versus "no algorithm use".
  Patients who fulfilled the above eligibility criteria will have their data collected and entered into the predictive algorithm.
Sampling Method: Non-Probability Sample
Enrollment: 689 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of predictive algorithm for acute appendicitis | 30 days
  Accuracy of predictive algorithm and accuracy of doctors with input from the algorithm in diagnosing acute appendicitis

CONTACTS AND LOCATIONS:
Overall Officials: Kee Yuan Ngiam, Dr, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.